CLINICAL TRIAL: NCT03016416
Title: The Influence of Rhythm, Cognitive Task and Physical Activity on the Cardiac Autonomic Nerve System in Chronic Stroke Patients and in a Control Group
Brief Title: The Influence of Rhythm, Cognitive Task and Physical Activity on the Cardiac ANS in Chronic Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Alon Erez, Doctor, Clalit Health Services
Other Study IDs: 0063-16-COM
Record Dates: First submitted 2016-12-25; First posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Unrecognized Condition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- chronic stroke patients: Participants for the study group will be recruited from the Clalit Health Services- Ben Yair Rehabilitation Center in Jaffa Israel.
- control group: The control group will be with equivalent age and lifestyle as the studt group. Participants for the control group will be recruited via solicitation adds at the Ben Yair Rehabilitation Center and at near-by clinics.

SUMMARY:
Autonomic dysfunction is a common complication of stroke that may lead to poor rehabilitation outcomes and to increase in mortality. The severity of the autonomic dysfunction can be measured in many ways, but the most common way is assessment of the sympathetic-parasympathetic equilibrium by heart rate variability analysis. It is known that the plasticity of the brain can influence the autonomic nerve system and that providing appropriate stimuli encourages these changes. It was found that stimulation of rhythm, stimulation of cognitive tasks and stimulation of activity, influence the autonomic nerve system in healthy subjects. Thus, we can ask if an integrated task (activity, cognitive, rhythm) may influence the autonomic nervous system and cause an increase in brain activity, therefore contributing to the rehabilitation of stroke patients. Taken together, the purpose of this study is to examine the influence of stimulation of rhythm, stimulation of cognition, stimulation of activity and combined stimulation, on the autonomic nerve system. This effect will be tested by measuring heart rate variability in chronic stroke patients and in a control group.

DETAILED DESCRIPTION:
background and Rationale: Autonomic dysfunction is a common complication of stroke that may lead to poor rehabilitation outcomes and to increase in mortality. Although this dysfunction is a common symptom of stroke, both in the acute phase and in the chronic phase, it is not a specific therapeutic target yet. The severity of the autonomic dysfunction can be measured in many ways, but the most common way is assessment of the sympathetic-parasympathetic equilibrium by heart rate variability analysis. It is known that the plasticity of the brain can influence the autonomic nerve system and that providing appropriate stimuli encourages these changes. It was found that stimulation of rhythm, stimulation of cognitive tasks (in particular, stimulation of executive functions) and stimulation of activity, influence the autonomic nerve system in healthy subjects. Thus, we can ask if an integrated task (activity, cognitive, rhythm) may influence the autonomic nervous system and cause an increase in brain activity, therefore contributing to the rehabilitation of stroke patients. Taken together, the purpose of this study is to examine the influence of stimulation of rapid or slow rhythm, stimulation of cognition by cognitive tasks, stimulation of activity by pedaling a fitness bike and combined stimulation, on the autonomic nerve system. This effect will be tested by measuring heart rate variability in chronic stroke patients and in a control group with equivalent age and lifestyle.

The Medical Device:

Heart rate and heart rate variability will be monitored by Polar RS800CX watch (PolarElectro OY, Kempele, Finland(. A transmitter placed on the patient's chest will collect the data. This data will be stored in the watch's computer and then analyzed in a specific Polar software (Polar Protrainer 5 inc.). An appropriate filtration will be made after a preliminary study. Pedaling capability, RPM, will be collected from cadence sensor with Bluetooth smart.

The Purpose of this Medical Research:

The purpose of this study is to examine the influence of stimulation of rapid or slow rhythm, stimulation of cognition by cognitive tasks, stimulation of activity by pedaling a fitness bike and combined stimulation, on the autonomic nerve system in chronic stroke patients and in a control group with equivalent age and lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be > 60 years, have Clalit health insurance, walking and Hebrew native speakers. Number of man and woman participating in the study will be equal.

Exclusion Criteria:

* Individuals with any of the following criteria will not participate in the study: participants with communication problems such as language, hearing or visual problems, recurrent strokes, cognitive deficiency (MoCA≤ 26) (Toglia et al., 2011), neglect by BIT - Star cancellation test (Wilsonet et al., 1987), patients with central or peripheral neurological problems, heart pacemaker and/or patients that use medications that effect the autonomic nerve system such asβ blockers, or use alcohol or drugs.
* Patients that suffer from background illness that can effect their ability to cycle such as knee OA.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The research will include two study groups, each with 16 participants. Participants in the study group will include 16 patients after first ischemic stroke, one sided, in the chronic phase.
  * Participants in the control group will include 16 healthy adults with equivalent age and lifestyle and without stroke history.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2017-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | 90 min
  Heart rate variability will be monitored by Polar RS800CX watch (PolarElectro OY, Kempele, Finland). A transmitter put on the patient's chest will collect the data. This data will be stored in the watch's computer and then analyzed in a specific Polar software (Polar Protrainer 5 inc.). An appropriate filtration will be made after a preliminary study.

SECONDARY OUTCOMES:
Pedaling capability | 25 min
  Pedaling capability, rpm, will be collected from cadence sensor with Bluetooth smart
Cognitive outcomes | 10 min task
  Cognitive outcomes will be evaluated by Digit Span, a sub section of Wechsler Adult Intelligence test (Choi et al., 2014).

IPD SHARING:
Plan to Share IPD: No